CLINICAL TRIAL: NCT02878824
Title: Role of Ethnicity and Environment on Regulation of Response Towards Sensory Stimulation in Children: A Neurophysiological Study
Brief Title: Role of Ethnicity and Environment on Regulation of Response Towards Sensory Stimulation in Children
Status: Completed | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, GOMEZ Ivan Neil Benitez, Mr., The Hong Kong Polytechnic University
Other Study IDs: HSEARS20150316001-01
Record Dates: First submitted 2016-08-15; First posted 2016-08-25 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Children; Behavior
Keywords: Neurophysiology; Autonomic; Sensory; Child; Ethnicity; Environment
MeSH Terms: conditions — Behavior | interventions — Ethnicity; Environment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- HK-Children: This is a group of typically-developing children ages 7-12 years old who are of Chinese ethnicity, born and raised in Hong Kong (n=32).
  Interventions: Other: Ethnicity
- FHK-Children: This is a group of typically-developing children ages 7-12 years old who are of Filipino ethnicity; either born, migrated and/or raised in Hong Kong (n=32).
  Interventions: Other: Ethnicity
- FU-Children: This is a group of typically-developing children ages 7-12 years old who are of Filipino ethnicity, born and raised in an urban area in the Philippines (n=32).
  Interventions: Other: Environment
- FR-Children: This is a group of typically-developing children ages 7-12 years old who are of Filipino ethnicity, born and raised in a rural area in the Philippines (n=32).
  Interventions: Other: Environment

INTERVENTIONS:
Other: Ethnicity — As mentioned by Goldberger and Veroff (1995) the concept of ethnicity is also associated with culture and is often used interchangeably with culture as well as with race. Ethnic differences are not necessarily inherited, but they are learned through constant exposure; however have strong genetic influences that explain consequent behavioural differences between different ethnic groups (Chudek & Henrich, 2011). An individual's genetic makeup greatly affects their behaviours (Klahr & Burt, 2014).
  In this study, we look at exposure to different ethnicity as exemplified by comparison between two groups of typically-developing children from different ethnicity (Chinese children in Hong Kong and Filipino Children in Hong Kong).
  Groups: FHK-Children; HK-Children
Other: Environment — The living environment has been implicated to have an effect on a person's psychological functioning (Rutter, Picker, Murray & Eaves, 2001) and eventually how behaviour is manifested. The proposed disparity or effects between urban and rural dwelling is built on research that looks at the restorative and calming features of the natural environment, as well as the chaotic organization of the living spaces in urban settings.
  Groups: FR-Children; FU-Children

SUMMARY:
Difference in autonomic nervous system processes across cultural and ethnic groups was suggested and autonomic regulation differentiation may occur even at an early age. However, the role of ethnicity and environment on regulation of response towards sensory stimulation in children is not well understood yet. This research aims to compare the autonomic activity at resting condition and toward a block of auditory stimulation between typically developing children from different countries and living environments. There will be two phases in this study. In Phase I, two groups of participants will be recruited: (a) 32 typically-developing Chinese children living in Hong Kong, (HK group) and (b) 32 typically developing Filipino children living in Hong Kong (Fil-HK group). In phase II, two groups of participants will be recruited: (a) 32 typically-developing Filipino children who are living at Urban area (PH-U group), and (b) 32 typically developing Filipino children who are living at Philippines-Rural area (PH-R group). Participants will be composed of males and females ages 7-12 years old, and without known history of developmental disabilities, medical history of cardiac or pulmonary problem, medical history of diabetes, or having any sensory deficits. Recruited participants will watch a silent movie, and listen to a block of sound. Autonomic activity (heart rate variability and electrodermal activity) will be measured and recorded using Polar H2 heart rate monitor and eSense skin response. Recordings will be screened for ectopic beats of HRV or bursts of EDA. The HRV and EDA signals will be processed by using aHRV and the eSense propriety software, respectively, and according to the standards of editing HRV and EDA artefacts. Autonomic activity (LF, HF and EDA) at resting condition, and hypothesis interaction between conditions (resting condition vs. auditory stimulation) and groups (HK group and PH-U group; Fil-HK group and PH-U group; PH-U group vs. PH-R group) will be tested with repeated measures of MANOVA. All significant levels will be set at p≤ 0.05. This study will increase the understanding on the role of culture and environment in the regulation of behaviour in auditory processing. The findings of this research may further shed light on the evaluation and treatment planning for children across and within cultures.

DETAILED DESCRIPTION:
Background: Difference in autonomic nervous system (ANS) processes across cultural and ethnic groups was suggested and autonomic regulation differentiation may occur even at an early age. However, the role of ethnicity and environment on regulation of response towards sensory stimulation in children is not well understood yet. This research aims to compare the autonomic activity at resting condition and toward a block of auditory stimulation between typically developing children from different countries and living environments and examine the role of environments and ethnicity on autonomic regulation.

Methods: Four groups of typically-developing participants will be recruited in this study: 1) Chinese children living in Hong Kong (n=32); Filipino children living in Hong Kong (32); Filipino children living in urban-Philippines (n=32); Filipino children living in urban-Philippines (n=32). Participants will be males (nm=16) and females (nf=16), ages 7-12 years old, and without known history of developmental disabilities, medical history of cardiac or pulmonary problem, medical history of diabetes, or having any sensory deficits. Recruited participants will watch a silent movie, and listen to a block of sound stimulus presentations. Autonomic activity (heart rate variability and electrodermal activity) will be measured and recorded using Polar H2 heart rate monitor and eSense GSR. Recordings will be screened for ectopic beats of HRV or bursts of EDA. The HRV and EDA signals will be processed by using aHRV and Ledalab software, respectively, and according to the standards of editing and analysing HRV and EDA artefacts. Autonomic activity (LF, HF and EDA) at experimental condition groups (HK group and PH-U group; Fil-HK group and PH-U group; PH-U group vs. PH-R group) will be tested with repeated measures of MANOVA. All significant levels will be set at a critical α=> .05.

Discussion: This study will increase the understanding on the role of culture and environment in the regulation of behaviour in auditory processing. The findings of this research may further shed light on the evaluation and treatment planning for children across and within cultures.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* 7-12 years old
* enrolled in primary school
* currently resides in the country/area in context
* for Hong Kong participants: Hong Kong-Chinese national
* for Philippine participants: born and living within the area in context

Exclusion Criteria:

* known history of developmental disabilities, medical history of cardiac or pulmonary problem, medical history of diabetes, or having any sensory deficits
* repeated a grade level
* multiracial parental background

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: For all participant groups, the recruited sample shall be males and females, aged 7-12 years old. Any participant with known history of developmental disabilities, medical history of cardiac or pulmonary problem, medical history of diabetes, or having any sensory deficits will be excluded. All participants will also be screened for past pertinent medical history for any maladaptive behaviour in sensory processing in daily living. Those showing definite problem in sensory processing will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2016-07; Primary Completion 2017-05 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | Day 1
  Heart rate variability (HRV) has been considered as a promising marker for autonomic activity, specifically of parasympathetic nervous system (PNS) activity (Task Force of the European Society of Cardiology and the North American Society for Pacing and Electrophysiology, 1996). Frequency domain analysis covers total power (0.0-0.5 Hz) in its raw and normalized units, low (LF; 0.04-0.15 Hz) and high (HF; 0.15-0.40 Hz) frequency components in its raw and normalized units. The normalized units of the LF will be used as representative of predominantly sympathetic modulation activity (SNS), while the normalized units of the HF will be used as representatives of parasympathetic modulation activity.
  Since HRV can measure both SNS and PNS simultaneously, this study will use HRV as one of the measurements. Nevertheless, it has been argued if the value of LF is a pure measure of SNS (Goldstein et al., 2011). Therefore, other than HRV, EDA will also be a supplementary measurement.
Electrodermal Activity | Day 1
  Electrodermal activity (EDA) is a valid measure of autonomic nervous system activity frequently used to index behavioural processes (Boucsein, Fowles, Grimnes, Ben-Shakhar & Roth, 2012). EDA is composed of a tonic and phasic drivers that reflect autonomic availability and response patterns respectively. Tonic EDA will be represented by the CDA.Tonic, which has been recommended to be the most accurate representation of the deconvoluted underlying skin conductance level within the specified block expressed in µS (Benedek & Kaernbach, 2010). To represent the sympathetic activity in the form of phasic skin conductance response, the CDA.SCR will computed. The CDA.SCR is considered as the average phasic driver within the specified response window initially set, and represents the phasic EDA most accurately expressed in units of µS (Benedek & Kaernbach, 2010).

SECONDARY OUTCOMES:
Sensory Behaviours: English and Chinese versions of the Sensory Profile | Day 1
  To measure the child's behavioural patterns in response to sensory stimulus in his daily activities, we will use the original Sensory Profile (Dunn, 1999) and Chinese Sensory Profile (Cheung & Siu, 2010). The original Sensory Profile which was developed and validated by Dunn (1999) is a 125 item questionnaire that is completed by the caregiver. The Chinese Sensory Profile was translated and validated by Cheung and Siu (2010) is a 100-item parent-report measure used among children and uses the same rating scale as with the original one. In this research, similar items from the original English version and Chinese versions of the Sensory Profile are identified and matched.
Temperament: English and Chinese versions of the Temperament in Middle Child Questionnaire and Early Adolescent Temperament Questionnaire | Day 1
  Temperament will be measured using the Temperament in Middle Childhood Questionnaire (TMCQ; Simonds & Rothbart, 2004; 2006) for 7-10 year old children; and the Early Adolescent Temperament Questionnaire (TMCQ; Ellis & Rothbart, 2001) for children 11-12 years old. TMCQ is a 157-item parent questionnaire, while EATQ s 65-item form with a scale; both are parent-rated measures of reactive and regulative temperament traits among children using a 5-point Likert scale (a range of "Almost always untrue-1" to "Almost always true-5") for each item. The original version was developed using the English language. The Chinese translation of TMCQ (Lay et al., 2004) and EATQ (Lay & Hsu, 2004) will be used Chinese-speaking participants.
Resilience: English and Chinese versions of the Child and Youth Resilience Measure | Day1
  The Child and Youth Resilience Measure [37] (CYRM) was established through a process of interviews with youth and adults in countries around the world was completed by the participants' parents. This research uses the 28-item (> 10 yrs. old) or 26 item (5-9 yrs. old) Person-Most-Knowledgeable questionnaire version, which was developed and validated by Ungar and Liebenberg [38]. While the CYRM is originally in English, a translated Chinese version was recommended and provided by the authors and was used among Chinese participants in this research. Parents rate each item with three possible response: "Yes," "Sometimes" or "No."

OTHER OUTCOMES:
Body-Mass Index | Day 1
  Body mass index (BMI) was ascertained through measurement of the participants' height (cm) and weight (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia YY Lai, PhD, Study Director — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided